CLINICAL TRIAL: NCT02297568
Title: Randomized Control Trial of Vitamin D Supplementation During Lactation on Vitamin D in Maternal Milk
Brief Title: Vitamin D Supplementation During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJVITD001
Record Dates: First submitted 2014-11-10; First posted 2014-11-21 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2015-07

CONDITIONS: Deficiency, Vitamin D
Keywords: Breast-fed infant; vitamin D supplementation; Lactation
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calciferol,1800 IU/d supplement (Active Comparator): The lactating mothers and their breastfed infants with maternal 25 Hydroxy-vitamin D (25OHD) levels of 10-30 ng/ml in third trimester were randomly assigned to 1,800 IU/d .
  Interventions: Drug: Calciferol
- Placebo (Placebo Comparator): The lactating mothers and their breastfed infants with maternal 25 Hydroxy-vitamin D (25OHD) levels of 10-30 ng/ml in third trimester were randomly assigned to receive placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Calciferol — Comparison 25OHD levels between calciferol and placebo
  Other Names: Vitamin D3
  Arms: Calciferol,1800 IU/d supplement
Drug: placebo
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled trial in Thai pregnancy is conducted. The study aims to determine whether vitamin D3 1,800 IU/d supplementation in lactating mother improves vitamin D status of breastfed infant.

DETAILED DESCRIPTION:
Vitamin D deficiency in pregnancy increases risk of gestational diabetes mellitus, pre-eclampsia, preterm birth, low birth weight and cesarean section. To against these adverse events, vitamin D supplementation in pregnancy and lactation is recommended, but dose ranges are varied. Then, this study is carried out in lactating mothers and their breastfed infants with maternal 25 Hydroxy-vitamin D (25OHD) levels of 10-30 ng/ml in third trimester. Subjects are divided into 2 groups, one is randomly assigned to 1,800 IU/d compared with maternal and infant controls receiving placebo. Maternal serum 25OHD and milk VitD will be measured by LC-MS/MS during lactation, and on cord blood at 6 weeks breastfed infants. This study is submitted for ethical consideration by relevant Ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Thai women and intends to deliver at Rajavithi Hospital
* Insufficient Vitamin D levels (25(OH)D < 30ng/ml)
* Gestational age at birth and no complications

Exclusion Criteria:

* Age < 18 years old
* Unintended to deliver at Rajavithi Hospital
* Insufficient Vitamin D levels (25(OH)D < 10ng/ml)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Comparison serum 25OHD levels from breastfed infants | 6 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sathit Niramitmahapanya, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand